CLINICAL TRIAL: NCT04186195
Title: Psychosocial and Socioeconomic Factors Affecting Glycemic Control in Children and Adolescents With Type 1 Diabetes Mellitus
Brief Title: Psychosocial Factors Affecting Glycemic Control in Children and Adolescents With Type 1 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: R19096
Record Dates: First submitted 2019-11-15; First posted 2019-12-04 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Glycemic control; Children; Psychosocial and socioeconomic factors
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diabetic children aged 1-16 years and their families: Diabetic children aged 1-16 years and their families. A child's disease duration must be over 1 year so that possible remission period is over.

SUMMARY:
The aim of the study is to research psychosocial and socioeconomic factors among families that might affect glycemic control in children and adolescent with type 1 diabetes mellitus. These factors might be: living conditions, structure of the family, socioeconomic status, divorces and parent's own glycemic control status (if parent's type 1 diabetes mellitus is present in the family).

DETAILED DESCRIPTION:
This study is going to clarify if there are some socioeconomical or psychosocial factors that might influence child's type 1 diabetes mellitus glycemic control. Study population consists of 300-350 diabetic children aged 1-16 years who have diabetic controls at Tampere University Hospital and their families. Required information is going to be collected with 2 questionnaires, wich families are kindly asked to fill in.

ELIGIBILITY:
Inclusion Criteria: Type 1 diabetic children aged 1-16 years and their parents. Patient's and parents' willingness to participate

Exclusion Criteria: Type 1 diabetes duration under 1 year. Difficulties to understand written finnish.

-

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Type 1 diabetic children aged 1-16 years followed at Tampere University Hospital and their parents . Child's disease duration minimum 1 year.
Sampling Method: Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Children's type 1 diabetes glycemic control | Through study completion, an average 5 years
  Socioeconomic and psychosocial factors affecting in type 1 diabetes glycemic status in children

SECONDARY OUTCOMES:
Parents' divorce rate | Through study completion, an average 5 years
  Frequency of parent's divorces in a family with a child with type 1 diabetes
Parent's type 1 diabetes glycemic status | Through study completion, an average 5 years
  Possible parent's own type 1 diabetes glycemic status correlation with a child's type 1 diabetes glycemic control

CONTACTS AND LOCATIONS:
Overall Officials: Marja-Terttu Saha, Principal Investigator — Tampere University
Locations (1):
- Tampere University Hospital, Tampere, Finland